CLINICAL TRIAL: NCT04997772
Title: Digital Health Platform Customized for Patients With Gaucher Disease
Status: Completed | Type: Observational
Sponsor: Shoshana Vilk (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor-Investigator, Shoshana Vilk, Prof. Shoshana Revel-Vilk, Shaare Zedek Medical Center
Organization: Shaare Zedek Medical Center (Other)
Other Study IDs: 0380-20-SZMC
Record Dates: First submitted 2021-07-28; First posted 2021-08-10 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Gaucher Disease; Patient Reported Outcome
Keywords: Gaucher Disease; Digital Health; Patient Reported Outcome
MeSH Terms: conditions — Gaucher Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Gaucher disease patients > 18 years old.
  Interventions: Device: Digital Gaucher Platform

INTERVENTIONS:
Device: Digital Gaucher Platform — Digital platform specified for Gaucher patients.

SUMMARY:
The entry of digitization into the world in recent years is helping the health care system to operate more efficiently than in the past and has increased the participation of patients and their families in managing their health care.

In a rare disease, such as Gaucher disease, patient involvement through digital technology is of great importance. Gaucher patients come for an inspection at the Gaucher unit once every six months. However, medical events, related and unrelated to Gaucher, may occur between these visits, some of which may be urgent. A digital Gaucher platform will allow for the updating of medical events occurring in the patient between these visits and will allow specialists to give up-to-date medical advice to the patient and the local doctor when needed. The Gaucha Digital Platform will provide digital tools (and applications) for self-management, monitoring and regular contact with the Gaucher Unit. The system will have an alert system that will allow accessible communication between the patient and the Gaucher unit. Moreover, patients with Gaucher disease need a lifelong commitment to their care; Enzyme replacement therapy (ERT) and substrate inhibitor therapy (SRT). When patients are monitored only once or twice a year, monitoring adherence to treatment may be a problem. Adherence to the treatment regimen is essential for achieving normalization. The system will have a system of reminders for treatment and a system for monitoring the receipt of treatment. The digital system will include quality of life questionnaires and pain questionnaires that will help to more comprehensively understand the patient's condition.

Finally, a Gaucher-adapted digital platform will ensure the collection of all relevant clinical data that is important for the treatment of a rare and multi-systemic disease such as Gaucher disease. A complete database will make it possible to create an anonymous database that will be used to find predictors of response to treatment, complications and commodities associated with Gaucher disease.

DETAILED DESCRIPTION:
With quality outcomes and value, the watchwords for health care in the 21st century, stakeholders around the globe are looking for innovative, cost-effective ways to deliver patient-centered, technology-enabled "smart" healthcare, both inside and outside hospital walls.The Digital transformation in health and care aims at supporting the management of health and well being while empowering the participation of people and facilitating the transformation of health and care services to more digitized, person-centered and community-based care models, thereby enabling better access to healthcare and the sustainability of health and care systems.

Globally, the investigators see also an increase in the desire of patients themselves to play an active role in their healthcare management. In rare disease, such as Gaucher Disease (GD), patient engagement through a combined digital technology may have added importance. It is recommended for patients with GD to be managed by a multidisciplinary team of experts having long-term experience with the diverse clinical manifestations and potential GD-related or unrelated co-morbidities, their follow-up visits at the center of excellence are usually on an annual or semi-annual basis. However, disease-related and un-related medical events may occur in-between these visits, some which may be emergent. A digital Gaucher platform will enable updating medical events occurring to the patient in-between these visits and enable the specialists to give updated medical consult to the patient and local physician when needed.

Furthermore, patients with GD need a life-long commitment to their therapy; enzyme replacement therapy (ERT) and substrate reduction therapy (SRT). The adherence to therapy regimen is essential to achieve normalization. When patients are followed only once-twice a year in a specialized clinic following the adherence to therapy might be a problem. A digital Gaucher-platform will provide digital tools (and applications) for self-management, adherence, and patient-reported outcome using a Gaucher-dedicated APP. Alert dashboard will be developed and installed for the health professionals in order to enable accessible communication between the patient and health professionals and be able to respond in a timely manner.

Patient-reported outcome (PRO) and Patient-reported outcome measures (PROMs) are increasingly important in research and clinical practice and to monitor the efficiency of health care services. The use of PROMs is fundamental to ensure that what matters to patients is captured in a valid, reliable, responsive, and feasible manner. A Digital Gaucher Platform can collect GD-specific PROMs.

Finally, a digital Gaucher platform will ensure capturing all relevant clinical data, full data files, and complete missing data, important endeavor for the treatment of the individual patients with a rare and multi-system disease such as GD. Data completion is essential for the development of a database, agnostic to pharma companies or ways of treatment, with high-quality real-time data. This database can then be used for big data analysis for finding predictors for GD-related complications and commodities.

ELIGIBILITY:
Inclusion Criteria:

1. All adults (>18 years, no age maximum) treated patients with GD will be eligible.
2. Signed informed consent.

Exclusion Criteria:

1. Patients without access to either computer or mobiles phone.
2. For this pilot study patients whose communication skills in Hebrew is not good enough to complete the study questionnaires and PROMs [the app platform will use a very simplified language, thus allowing patients with limited Hebrew to use the app] *for future use/study the platform will be translated to other languages, as needed.

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Gaucher disease patients above the age of 18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Rate of satisfaction from Gaucher treatment at baseline compared to the end of study | 12 months
  GD-PROMs

SECONDARY OUTCOMES:
Adherence to treatment based on participant reports in the App | 12 months
  participants report in the app
Achievement of treatment goals based on Gaucher consensus paper | 12 months
  Gaucher consensus paper

CONTACTS AND LOCATIONS:
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No